CLINICAL TRIAL: NCT01815411
Title: Effect of the Mushroom Extract Andosan on Symptoms and Inflammatory Parameters in Patients With Rheumatoid Arthritis (RA)
Brief Title: Effect of Andosan in Patients With Rheumatoid Arthritis
Acronym: Andosan-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egil Johnson (Other)
Collaborators: ImmunoPharma AS (Industry)
Responsible Party: Sponsor-Investigator, Egil Johnson, consultant, professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012/1962; Egil Johnson (Other: Dep. of gastroenterological- and pediatric surgery, Ulleval)
Record Dates: First submitted 2013-03-14; First posted 2013-03-21 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; symptom score; fatigue; life quality; cytokines; mRNA expression; Quality of Life; Signs and Symptoms; Indication for Modification of Patient Physical Status
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mushroom extract (Experimental): The patients are given the mushroom extract (Andosan) in doses 30 mlx2 per day for 1 days. The experimental group is selected by randomisation.
  Interventions: Dietary Supplement: Mushroom extract
- Control group (No Intervention): The control group is selected by randomisation.

INTERVENTIONS:
Dietary Supplement: Mushroom extract — The mushroom extract (Andosan) is given orally in doses 30 m x 2 daily for 21 days
  Arms: Mushroom extract

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic, autoimmune inflammatory disease that leads to significant pain, joint destruction and functional decline, and has a substantial economic impact both for sufferers and society. Although the etiology of RA is unknown, it is generally accepted that it arises from an interplay of genetic predisposition (in particular, HLA-DR allele subtypes and specific gene polymorphisms), immunological deregulation (e. g. autoantibody production), and environmental factors. The prevalence and incidence of RA in Norway is estimated to 0,4-0,5 % and 0,020-0,025 %, respectively, and incidence rates are 2-4-fold higher in women. Synovitis and bone resorption are key pathogenetic factors in RA and these patients have elevated cytokine levels in joints and blood (i.e. TNF, IL-1, IL-6). RA is also associated with significant comorbidity; the most important is premature cardiovascular disease that significantly contributes to increased mortality. Compared with the general population, mortality in RA is from 1,57-2,0-fold higher in Norway and Sweden, and their mean life expectancy is reduced by an average of 5-10 years. Medical treatment of RA consists of nonsteroidal anti-inflammatory drugs, systemic glucocorticosteroids, traditional disease modifying antirheumatic drugs (including methotrexate) and biologic therapies (including anti-tumor necrosis factor (TNF) α, anti-IL 6 and anti-CD20 therapy). Also, a considerable portion of the patients are in need of joint replacement surgery and in need of rehabilitation.

However, the treatment opportunities are still not optimal. In a large proportion of the patients, full control of the disease is not possible due to limited effect of available therapies and/or intolerance to these therapies. Therefore, there is a huge need to find new therapeutic alternatives to treat RA.

Since studies on healthy volunteers and IBD-patients support that the mushroom extract AndoSanTM exert an anti-inflammatory effect in vivo, the investigators wanted to examine in a pilot study whether this effect also was evident in patients with RA. A potential anti-inflammatory effect could prove beneficial in these seriously ill patients, who accordingly could experience less side effects (edema, granulocytopenia, diminished tissue repair) due to potential reduction number and dose of disease modifying drugs.

DETAILED DESCRIPTION:
Main aim: Examine whether daily oral ingestion of a immunomodulatory mushroom extract (AndoSanTM) leads to a clinical, biochemical and genetical improvement in RA. The experiment will be carried out for 21 days in 15 eligible RA patients. In order to increase the scientific value of the project we will use, a as far as possible, an age matched control group of RA patients with steady medication and no intervention. The control group of 10-15 patients will be answering the same questionnaires and give the same samples of blood and feces.

Partial aims: To compare prior to (day 0) and after (day 21) daily (30 ml x 2) ingestion of Andosan the effect of this therapy on:

* general blood samples (leucocytes, CRP, liver and renal function tests), including erythrocyte sedimentation rate (SR) and pentraxin 3 (PTX3)
* level of blood cytokines and analytes (IL-1α/-1ra/-2/-4/-5/-6/-7/-8/-9/-10/-12(p70)/-13/-15/ 17,G-CSF,GM-CSF,MCP-1,MIP-1ß/-1α,IFNγ,TNFα and basic FGF, eotaxin, PDGF-BB, RANTES,VEGF;27-plex) -level of inflammatory marker calprotectin in feces and blood in patients
* genetic expression in blood leukocytes (microarray) -number of swollen and tender joints, morning stiffness, Disease activity score 28 calculated by ESR (DAS28-ESR), RA impact of disease score (RAID), Health Assessment Questionnaire (HAQ), visual analogue scale (VAS) for patient's and physician's global assessment of disease activity, life quality (SF-36 version 2), fatigue score.

Partial aims: To compare prior to (day 0) and after (day 21) daily (30 ml x 2) ingestion of Andosan the effect of this therapy on:

* general blood samples (leucocytes, CRP, liver and renal function tests), including erythrocyte sedimentation rate (SR) and pentraxin 3 (PTX3)
* level of blood cytokines and analytes (IL-1α/-1ra/-2/-4/-5/-6/-7/-8/-9/-10/-12(p70)/-13/-15/ 17,G-CSF,GM-CSF,MCP-1,MIP-1ß/-1α,IFNγ,TNFα and basic FGF, eotaxin, PDGF-BB, RANTES,VEGF;27-plex) -level of inflammatory marker calprotectin in feces and blood in patients
* genetic expression in blood leukocytes (microarray) -number of swollen and tender joints, morning stiffness, Disease activity score 28 calculated by ESR (DAS28-ESR), RA impact of disease score (RAID), Health Assessment Questionnaire (HAQ), visual analogue scale (VAS) for patient's and physician's global assessment of disease activity, life quality (SF-36 version 2), fatigue score.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Able and willing to give written informed consent, and to comply with the requirements of the study protocol.
* Fulfilling the ACR 1987 revised diagnostic criteria for the diagnosis rheumatoid arthritis.
* Moderate disease activity based on the clinical evaluation including DAS28-ESR (DAS28 3.2-5.1) [11, 12].
* Stable medication by disease modifying drugs (DMARDs) and systemic glucocorticosteroids for 3 months prior to the inclusion.

Exclusion Criteria:

* Lack of cooperativity.
* Clinically significant chronic infection, including positive serology for hepatitis B or C, history of positive HIV status.
* Acute significant infection during the last 3 weeks before the inclusion. Surgery during the last 4 weeks before the inclusion, and during the study period.
* Clinically significant malignancy .
* Drug addiction
* Any inflammatory disease of permanence not related to RA.
* Use of prednisolone >7,5 mg daily for 1 month prior to the inclusion.
* Use of biologic treatment including antibodies to cytokines and their receptors for 6 weeks prior to the inclusion.
* Use of intramuscular, intra-articular or intravenous injections of corticosteroids during or within 4 weeks prior to inclusion in the trial.
* Vaccination during the trial.
* Pregnancy or breast-feeding.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Symptom score | The duration of the experiment is 3 weeks (21 days)
  The symptom score will be registered at day 1 prior to the patients are given Andosan for 21 days, and at day 21 after the patients have consumed Andosan daily for 21 days.

SECONDARY OUTCOMES:
Cytokine levels in harvested blood from the patients | The duration of the experiment is 3 weeks (21 days)
  Cytokine levels will be measured at day 1 prior to ingestion of Andosan and at day 21 after 21 days of Andosan consumption.

OTHER OUTCOMES:
Life quality (SF-36) | The duration of the experiment is 3 weeks (21 days)
  The patients will be registerd for life quality prior to ingestion of Andosan at day 1 and at day 21 after daily ingestion of Andosan for 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Egil Johnson, Md, PhD, Principal Investigator — Dep. of gastric- and pediatric surgery, Oslo University Hospital, Ulleval, Kirkeveien 166, 0407 Oslo
Locations (1):
- Lillehammer Hospital for Rheumatic Diseases, Lillehammer, Norway

REFERENCES:
- [Background] Johnson E, Forland DT, Hetland G, Saetre L, Olstad OK, Lyberg T. Effect of AndoSan on expression of adhesion molecules and production of reactive oxygen species in human monocytes and granulocytes in vivo. Scand J Gastroenterol. 2012 Sep;47(8-9):984-92. doi: 10.3109/00365521.2012.660544. Epub 2012 May 8. PMID 22564240
- [Background] Forland DT, Johnson E, Saetre L, Lyberg T, Lygren I, Hetland G. Effect of an extract based on the medicinal mushroom Agaricus blazei Murill on expression of cytokines and calprotectin in patients with ulcerative colitis and Crohn's disease. Scand J Immunol. 2011 Jan;73(1):66-75. doi: 10.1111/j.1365-3083.2010.02477.x. PMID 21129005
- [Background] Hetland G, Johnson E, Lyberg T, Kvalheim G. The Mushroom Agaricus blazei Murill Elicits Medicinal Effects on Tumor, Infection, Allergy, and Inflammation through Its Modulation of Innate Immunity and Amelioration of Th1/Th2 Imbalance and Inflammation. Adv Pharmacol Sci. 2011;2011:157015. doi: 10.1155/2011/157015. Epub 2011 Sep 6. PMID 21912538